CLINICAL TRIAL: NCT01934725
Title: Searching for Explanations for Cryptogenic Stroke in the Young: Revealing the Etiology, Triggers, and Outcome (SECRETO)
Brief Title: Searching for Explanations for Cryptogenic Stroke in the Young: Revealing the Etiology, Triggers, and Outcome
Acronym: SECRETO
Status: Active, not recruiting | Type: Observational
Sponsor: SECRETO Study Consortium (Other)
Collaborators: Finnish Medical Foundation (Network); Academy of Finland (Other); Hospital District of Helsinki and Uusimaa (Other); Hospital District of Southwestern Finland (Other); Pirkanmaa Hospital District (Unknown); Hospital District of North Ostrobothnia (Unknown); Northern Savo Hospital District (Other); Sahlgrenska University Hospital (Other); Sigrid Jusélius Foundation (Other)
Responsible Party: Principal Investigator, Jukka Putaala, Associate Prof., MD, PhD, MSc, SECRETO Study Consortium
Other Study IDs: SECRETO
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Brain Infarction; Ischemic Stroke; Thrombosis; Foramen Ovale, Patent
Keywords: Ischemic Stroke; Brain Infarction; Patent Foramen Ovale; Stroke in the Young; Myocardial Infarction; Cerebral Venous Thrombosis; Pulmonary Embolism; Deep Vein Thrombosis; Subarachnoid Hemorrhage; Prognosis; Databases, Genetic
MeSH Terms: conditions — Brain Infarction; Ischemic Stroke; Thrombosis; Foramen Ovale, Patent; Myocardial Infarction; Intracranial Thrombosis; Pulmonary Embolism; Venous Thrombosis; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients at baseline:
  4 x 2.7 mL sodium citrate tube, aliquoted in 10 x 300 µL cryovials; 1 x 5 mL PPACK sodium citrate tube, aliquoted in 5 x 300 µL cryovials; 1 x 8 mL serum tube, aliquoted in 5 x 300 µL cryovials; 1 x 9 mL EDTA tube #1, aliquoted in 10 x 300 µL cryovials; 1 x 9 mL EDTA tube #2, full blood for DNA extraction.
  Patients at 3-month visit (fasting): 4 x 2.7 mL sodium citrate tube, aliquoted in 10 x 300 µL cryovials; 1 x 5 mL PPACK sodium citrate tube, aliquoted in 5 x 300 µL cryovials; 1 x 8 mL serum tube, aliquoted in 5 x 300 µL cryovials; 1 x 9 mL EDTA tube, aliquoted in 10 x 300 µL cryovials.
  Control subjects:
  4 x 2.7 mL sodium citrate tube, aliquoted in 10 x 300 µL cryovials; 1 x 5 mL PPACK sodium citrate tube, aliquoted in 5 x 300 µL cryovials; 1 x 8 mL serum tube, aliquoted in 5 x 300 µL cryovials; 1 x 9 mL EDTA tube #1, aliquoted in 10 x 300 µL cryovials; 1 x 9 mL EDTA tube #2, full blood for DNA extraction.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients w/ cryptogenic ischemic stroke: Patients aged 15 to 49 years with unexplained first-ever ischemic stroke
- Stroke-free control subjects: Stroke-free subjects age- and gender-matched to patients

SUMMARY:
BACKGROUND: In industrialized countries a considerable and increasing proportion of strokes occur at younger ages. Stroke at young age causes marked disability at worst and thus long-standing socioeconomic consequences and exposes survivors for 4-fold risk of premature death compared with background population. Up to 50% of young patients with ischemic stroke remain without definitive etiology for their disease despite extensive modern diagnostic work-up (i.e. cryptogenic stroke). The group of cryptogenic strokes includes those with patent foramen ovale (PFO) or other abnormalities in the atrial septum in the heart as the only or concomitant finding. Population prevalence of PFO is high, 25%, and the mechanisms how PFO would be associated causally with ischemic stroke remain to be clarified. Moreover, there are only scarce data on clinical outcome, long-term risk of new vascular events, and prevention of such events in these patients.

DESIGN: Searching for Explanations for Cryptogenic Stroke in the Young: Revealing the Etiology, Triggers, and Outcome (SECRETO) is an international prospective multicenter case-control study of young adults (age 18-49) presenting with an imaging-positive first-ever ischemic stroke of undetermined etiology (aim N=2000). Patients are included after standardized diagnostic procedures (brain MRI, imaging of intracranial and extracranial vessels, cardiac imaging, and screening for coagulopathies) and age- and sex-matched to healthy controls in a 1:1 fashion. Up to 45 study sites worldwide will be needed to recruit the planned participant population during a 3-year period. Neurovascular imaging and echocardiography studies, and ECGs will be read centrally.

AIMS: SECRETO involves five principal fields of investigation: (1) Stroke triggers and clinical risk factors; (2) Long-term prognosis (new vascular events, functional and psychosocial outcomes); (3) Abnormalities of thrombosis and hemostasis; (4) Biomarkers of e.g. inflammation, atherogenesis, endothelial function, thrombosis, platelet activation, and hemodynamic stress to characterize postulated cryptogenic stroke mechanisms; and (5) genetic study, including genome-wide association and candidate gene studies as well as next-generation sequencing approach. All analyses consider cardiac functional and interatrial structural properties as a possible mediator. Furthermore, SECRETO Family Study (substudy) aims at collecting extensive family history of thrombotic events from informative patients being screened for SECRETO main study and collect genetic samples from all consenting family members for whole-genome sequencing.

SIGNIFICANCE: SECRETO will provide novel information on clinical and subclinical risk factors, both transient and chronic, predisposing to cryptogenic ischemic stroke in young adults. This study also reveals long-term prognosis of this understudied patient population and may discover new genetic background underlying the disease mechanism and provide potential targets for drug development.

ELIGIBILITY:
PATIENTS:

Inclusion Criteria:

1. Age 18 to 49 at stroke onset
2. Patient hospitalized due to first-ever imaging-positive ischemic stroke of undetermined etiology after complete timely diagnostic testing.

Exclusion Criteria:

1. Baseline mandatory tests not obtained in the first week following stroke onset, including:

   * Brain MRI
   * Routine blood tests, including complete blood count, CRP, fasting glucose, creatinine, aPTT, INR, total cholesterol, LDL-cholesterol, HDL-cholesterol, HbA1C, hemoglobin electrophoresis in individuals of African origin
2. Other baseline mandatory tests not obtained within the first two weeks following stroke onset, including:

   * Imaging of cervicocephalic arteries by CTA, MRA, or DSA
   * Transesophageal (highly recommended) or transthoracic echocardiography
   * 24-hour Holter monitoring or continuous in-hospital ECG monitoring with automated arrhythmia detection for at least 24 hours
   * Screening for thrombophilia, including antiphospholipid antibodies and other coagulopathies (any abnormal finding must be retested at mandatory 3-month follow-up visit >12 weeks from initial testing or >4 weeks after cessation of anticoagulation at any later time point); mandatory tests include anticardiolipin antibodies, lupus anticoagulant, anti-β2-glycoprotein antibodies, factor V mutation (or aPC resistency ruled out), factor II mutation, homocysteine, antithrombin III, protein C, and protein S
3. No evidence of current brain ischemia
4. Current stroke due to cerebral venous thrombosis or as a complication of subarachnoid hemorrhage, angiography, or cardiac surgery
5. Patient otherwise not eligible for the study or adherent for follow-up (eg nonresident) or has concurrent disease affecting outcome (eg multiple sclerosis, cancer)
6. Informed consent not obtained from the patient or a proxy.

CONTROL SUBJECTS:

Inclusion Criteria:

1. Age 18 to 49 years
2. Absence of prior ischemic stroke as ascertained using the Questionnaire for Verifying Stroke-Free Status

Exclusion Criterion:

1. Informed consent not obtained

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Patients aged 18 to 49 hospitalized due to first-ever imaging-positive ischemic stroke of undetermined etiology;
  2. Age-, gender- and race-ethnicity-matched stroke-free control subjects
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Nonfatal or fatal recurrent ischemic cerebrovascular event | 10 years
  Ischemic stroke or transient ischemic attack

SECONDARY OUTCOMES:
Composite of noncerebrovascular arterial or venous thrombotic events, or cerebral venous thrombosis | 10 years
Death from any cause | 10 years
New-onset atrial fibrillation | 10 years

OTHER OUTCOMES:
Modified Rankin Scale | 10 years
  Functional outcome will be assessed with modified Rankin Scale at mandatory 3-month visit and at annual follow-up contacts from year 1 to year 10.
Vocational outcome | 10 years
  Vocational status will be assessed at each follow-up contact with Poststroke Working Activity Questionnaire and a set of questions designed for the study.
Cognitive outcome | 3 months
  Cognition will be assessed at mandatory 3-month follow-up visit (Montreal Cognitive Assessment).
Anxiety and depression | 10 years
  Poststroke anxiety and depression will be evaluated at 3-month visit, 1-year, 5-year, and 10-year follow-up contacts with Hospital Anxiety and Depression Scale.
Quality of life | 10 years
  Quality of life will be assessed at 3-month visit, 1-year, 5-year, and 10-year follow-up contacts with EuroQol questionnaire.
Caregiver burden | 3 months
  Poststroke burden to caregiver will be assessed at 3-month visit with Expanded Caregiver Strain Index Questionnaire.
Barthel Index | 10 years
  Functional outcome will be assessed with Barthel Index at mandatory 3-month visit and at annual follow-up contacts from year 1 to year 10.

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Putaala, A/Prof., Principal Investigator — Helsinki University Central Hospital; Steven Kittner, Prof., Principal Investigator — University of Maryland Hospital
Locations (19):
- Tartu University Hospital, Tartu, Estonia
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- Ernst-Moritz-Arndt University Medicine, Greifswald, Germany
- "Attikon" Hospital, University of Athens, School of Medicine, Athens, Greece
- Italy (2):
  - University of Brescia, Brescia
  - Arcispedale S. Maria Nuova, Reggio Emilia
- Vilnius University Hospital Santariskiu klinikos, Vilnius, Lithuania
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Haukeland University Hospital, Bergen, Norway
- Hospital Santa Maria, Lisbon, Portugal
- Torrecárdenas University Hospital, Almería, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Istanbul University Istanbul Faculty of Medecine, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Peterborough City Hospital, Peterborough
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Putaala J, Martinez-Majander N, Leppert M, Tulkki L, Pirinen J, Tolppanen H, Sarkanen T, Virtanen M, Jaakonmaki N, Jakala P, Hedman M, Redfors P, Bech-Hanssen O, Junttola U, Huhtakangas J, Ylikotila P, Lautamaki R, Schminke U, von Sarnowski B, Busch R, Yesilot N, Sezgin M, Waje-Andreassen U, Saeed S, Fonseca AC, Paula A, Amaya Pascasio L, Martinez-Sanchez P, Korv J, Muda P, Ferdinand P, Oxley C, Zakarkaite D, Ryliskiene K, Pezzini A, Lombardi CM, Licenik R, Zedde M, Grimaldi T, Tsivgoulis G, Sinisalo J, Gerdts E, Tatlisumak T; SECRETO Study Group. Burden of Modifiable Risk Factors in Young-Onset Cryptogenic Ischemic Stroke by High-Risk Patent Foramen Ovale. Stroke. 2025 Jun;56(6):1428-1440. doi: 10.1161/STROKEAHA.124.049855. Epub 2025 Apr 17. PMID 40242852
- [Derived] Kutal S, Tulkki LJ, Sarkanen T, Redfors P, Jood K, Nordanstig A, Yesilot N, Sezgin M, Ylikotila P, Zedde M, Junttola U, Fromm A, Ryliskiene K, Licenik R, Ferdinand P, Jatuzis D, Korv L, Korv J, Pezzini A, Sinisalo J, Lehto M, Gerdts E, Autere J, Fonseca AC, Waje-Andreassen U, Von Sarnowski B, Sairanen T, Tatlisumak T, Huhtakangas J, Jakala P, Putaala J, Martinez-Majander N. Association Between Self-Perceived Stress and Cryptogenic Ischemic Stroke in Young Adults: A Case-Control Study. Neurology. 2025 Mar 25;104(6):e213369. doi: 10.1212/WNL.0000000000213369. Epub 2025 Mar 5. PMID 40043226
- [Derived] Sindre RB, Gerdts E, Putaala J, Grymyr LMD, Midtbo H, Almeida AG, Bech-Hanssen O, Busch R, Eilertsen RK, Fonseca AC, Hedman M, Huhtakangas J, Jakala P, Lautamaki R, Lehto M, Martinez-Majander N, Redfors P, Sarkanen T, von Sarnowski B, Sinisalo J, Virtanen M, Waje-Andreassen U, Yesilot N, Ylikotila P, Cramariuc D. Association of Left Atrial Stiffness With Risk of Cryptogenic Ischemic Stroke in Young Adults. JACC Adv. 2024 Mar 14;3(4):100903. doi: 10.1016/j.jacadv.2024.100903. eCollection 2024 Apr. PMID 38939654
- [Derived] Zedde M, Grisendi I, Assenza F, Napoli M, Moratti C, Bonacini L, Di Cecco G, D'Aniello S, Pavone C, Merlino G, Putaala J, Valzania F, Pascarella R. The Prepetrous Segment of the Internal Carotid Artery as a Neglected Site of Symptomatic Atherosclerosis: A Single-Center Series. J Clin Med. 2024 Mar 15;13(6):1696. doi: 10.3390/jcm13061696. PMID 38541922
- [Derived] Tulkki L, Martinez-Majander N, Haapalahti P, Tolppanen H, Sinisalo J, Repo O, Sarkanen T, Numminen H, Ryodi E, Ylikotila P, Roine RO, Lautamaki R, Saraste A, Miettinen T, Autere J, Jakala P, Hedman M, Huhtakangas J, Junttola U, Putaala J, Pirinen J; SECRETO Study Group. 24-hour ambulatory blood pressure and cryptogenic ischemic stroke in young adults. Ann Med. 2023 Dec;55(1):2203513. doi: 10.1080/07853890.2023.2203513. PMID 37086083
- [Derived] Kuusisto JK, Poyhonen PAK, Pirinen J, Lehmonen LJ, Raty HP, Martinez-Majander N, Putaala J, Sinisalo J, Jarvinen V. Revisiting left atrial volumetry by magnetic resonance imaging: the role of atrial shape and 3D angle between left ventricular and left atrial axis. BMC Med Imaging. 2021 Nov 9;21(1):167. doi: 10.1186/s12880-021-00701-5. PMID 34753444
- [Derived] Poyhonen P, Kuusisto J, Pirinen J, Raty H, Lehmonen L, Paakkanen R, Martinez-Majander N, Gerdts E, Putaala J, Sinisalo J, Jarvinen V. Right atrium and cryptogenic ischaemic stroke in the young: a case-control study. Open Heart. 2021 May;8(1):e001596. doi: 10.1136/openhrt-2021-001596. PMID 34006504
- [Derived] Poyhonen P, Kuusisto J, Jarvinen V, Pirinen J, Raty H, Lehmonen L, Paakkanen R, Martinez-Majander N, Putaala J, Sinisalo J. Left ventricular non-compaction as a potential source for cryptogenic ischemic stroke in the young: A case-control study. PLoS One. 2020 Aug 14;15(8):e0237228. doi: 10.1371/journal.pone.0237228. eCollection 2020. PMID 32797064
- [Derived] Pirinen J, Jarvinen V, Martinez-Majander N, Sinisalo J, Poyhonen P, Putaala J. Left Atrial Dynamics Is Altered in Young Adults With Cryptogenic Ischemic Stroke: A Case-Control Study Utilizing Advanced Echocardiography. J Am Heart Assoc. 2020 Apr 7;9(7):e014578. doi: 10.1161/JAHA.119.014578. Epub 2020 Mar 25. PMID 32208831
- [Derived] Martinez Majander N, Sinisalo J, Sundararajan S, Strbian D, Putaala J. Cryptic Loss of Consciousness in a 36-Year-Old Woman. Stroke. 2015 Jul;46(7):e164-6. doi: 10.1161/STROKEAHA.115.009405. Epub 2015 May 12. No abstract available. PMID 25967578
- See also: Study website — http://www.secretostudy.net